CLINICAL TRIAL: NCT06811337
Title: A 36 - Month Randomized Controlled Trial Comparing the Marginal Bone Changes Surrounding Dental Implants Placed With Open Versus Closed Sinus Elevation and Allogenic Bone Grafting.
Brief Title: Marginal Bone Changes Around Dental Implant Placed With Open vs. Closed Sinus Elevation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Misr International University (Other)
Collaborators: Suez Canal University (Other)
Responsible Party: Principal Investigator, Hebatallah Abdo's Elsaid Mattar, Assistant Lecturer - Oral & Maxillofacial Surgery Department, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021/419
Record Dates: First submitted 2025-01-19; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Marginal Bone Levels; Open Sinus Elevation; Closed Sinus Elevation
Keywords: Dental Implants; Bone Loss; Maxillary Sinus Floor Augmentation.; Bone-Implant Interface; Bone Resorption,
MeSH Terms: conditions — Bone Diseases, Metabolic; Bone Resorption

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lateral Sinus Elevation (Experimental)
  Interventions: Procedure: Open Sinus Elevation
- Transcrestal Sinus Elevation (Active Comparator)
  Interventions: Procedure: Closed Sinus Elevation

INTERVENTIONS:
Procedure: Open Sinus Elevation — Open Sinus Elevation
  Arms: Lateral Sinus Elevation
Procedure: Closed Sinus Elevation — Closed Sinus Elevation
  Arms: Transcrestal Sinus Elevation

SUMMARY:
Background: In cases with atrophic posterior maxilla, sinus elevation techniques are essential for a successful implant placement. The optimal strategy for treating pneumatized maxillary sinus in terms of dental implant insertion and surrounding bone stability has been a scientific conundrum for many years. The objective of this study was to evaluate and contrast the long-term marginal bone alterations around dental implants that were positioned utilizing transcrestal (closed) versus lateral (open) sinus elevation procedures.

Material and methods:

Fifty six dental implants were inserted for patients with inadequate residual bone height due to maxillary sinus pneumatization after receiving approval from Suez Canal University's ethics council. Depending on the method, these patients were randomly assigned to one of two groups: the test group, which received the closed sinus elevation, or the control group, which received the open sinus elevation.Allogenic bone grafting was used to treat the elevated sinuses in both groups.The mesial and distal marginal bone loss for these dental implants was evaluated over a 12-month period following surgery using a standardized digital periapical radiography and the Cliniview Software to measure radiographic bone alterations.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have at least one missing posterior maxillary tooth with sound adjacent teeth.
* Adults above the age of 18.
* Bone height from 4mm to 7mm under the maxillary sinus assessed in CBCT.
* Good oral hygiene.
* Patient accepts to sign an informed consent.

Exclusion Criteria:

* Smokers (more than 10 cigarettes per day).
* Medically compromised patients.
* Patients with active infection related at the site of implant/bone graft placement.
* Patients with untreated active periodontal diseases.
* Patients with parafunctional habits.
* Acute or chronic sinusitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Mesial and Distal marginal bone loss | 3 years
  Utilizing A standardized digital periapical radiography, and the Cliniview Software to measure radiographic bone changes mesially and distally to 56 implants placed after sinus elevation in the posterior maxilla.

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Ismailia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No